CLINICAL TRIAL: NCT00790257
Title: A Monocentre Phase 1 Trial to Assess a Monolayer Cellular Device in the Treatment of Type 1 Diabetes
Brief Title: Safety and Efficacy Study of Encapsulated Human Islets Allotransplantation to Treat Type 1 Diabetes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-HIA-002
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Islets transplantation; Encapsulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Monolayer Cellular Device (Experimental): Encapsulated human islets allotransplantation transplanted in subcutaneous tissue in Type 1 diabetes patient
  Interventions: Device: Encapsulated human islets in a "Monolayer Cellular Device"

INTERVENTIONS:
Device: Encapsulated human islets in a "Monolayer Cellular Device" — The product consists of isolated allogeneic human islets of Langerhans formulated in a serum-free transplant media. The islets will be encapsulated in an alginate-based "Monolayer Cellular Device".
  One device will be transplanted subcutaneously and corresponds to a patch of 1-3cm². One Device per patient. No Retransplantation.
  Other Names: MCD

SUMMARY:
In view to avoid immunosuppression, the investigators are submitting a Phase 1 clinical trial protocol testing the safety and the efficacy of encapsulated human islets in a "Monolayer Cellular Device" for allogeneic islets transplantation in Type 1 diabetic patients performed at the University clinical hospital Saint-Luc, Brussels. Encapsulated human islets will be transplanted in the subcutaneous tissue as "safety procedure" for patients.

This protocol (single center trial) is designed as a limited series of islets transplants for 15 Type 1 diabetic adult subjects.

DETAILED DESCRIPTION:
The need for chronic immunosuppressive therapy is paralleled by the occurrence of undesirable side effects in islets transplantation as well as whole pancreas transplantation. Several complications are associated with the administration of standard immunosuppressive agents (based on use of Sirolimus and Tacrolimus for example) used for human islets allotransplantation.

The herein presented protocol is a Phase 1 pilot study. This will be a single center clinical study. Study will be divided in 2 Phases.

* Phase 1A: T1DM patients, already transplanted with an organ (kidney, heart, liver or totally unfunctioning primary whole vascularized pancreas) and under immunosuppression, will receive the "Monolayer Cellular Device" in subcutaneous tissue in view to assess the capacity of encapsulated human islets to secrete insulin without immunological reaction.
* Phase 1B: T1DM patients will receive the "Monolayer Cellular Device" in subcutaneous tissue without immunosuppression in view to assess the biocompatibility of the device.

This protocol is designed as a limited series of islets transplants for 15 Type 1 diabetic adult subjects. In both Pase 1A/1B: Vascularized pancreas transplantation cannot be proposed, for these patients, following vascular disease, the older age, psychological reasons. Phase 1A consists in the transplantation of encapsulated human islets in Type 1 diabetic patients already transplanted with primary vascularized organ and under immunosuppression therapy.

Phase 1B consists in the transplantation of encapsulated human islets in Type 1 diabetic patients who cannot be eligible for whole vascularized pancreas transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1A:

  1. Male or female patients, of 30 to 80 years of age, C-peptide-negative;
  2. Patient must have signed the Patient Informed Consent Form;
  3. Type 1 diabetic (T1DM) patients insulin-dependent;
  4. T1DM patients already transplanted with a kidney graft and already on immunosuppressive therapy;
  5. T1DM patients already transplanted with a vascularized pancreas, already on immunosuppressive therapy, but with TOTAL dysfunction of the graft;
  6. T1DM patients already transplanted with a liver graft and already on immunosuppressive therapy;
  7. T1DM patients already transplanted with a heart or lung graft and already on immunosuppressive therapy;
  8. T1DM patients eligible for simultaneous transplantation with kidney and encapsulated human islets;
  9. Donor-Recipient ABO blood group compatibility;
  10. Donor- Recipient HLA compatibility.
* Phase 1B:

  1. Male or female patients, of 30 to 80 years of age, C-peptide-negative;
  2. Patient must have signed the Patient Informed Consent Form;
  3. T1DM patients without any immunosuppression who cannot be transplanted with vascularized pancreas (vascular complication, psychological reasons,...). The main objective is to restore a residual insulin secretion to stabilize the diabetes (reduction of hypoglycaemia,…);
  4. Donor-Recipient ABO blood group compatibility;
  5. Donor- Recipient HLA compatibility.

Exclusion Criteria:

* RECIPIENT EXCLUSION CRITERIA FOR PHASE 1A/B:

  1. Patient is pregnant or breastfeeding.
  2. Patient has a positive T-cell crossmatch on the most recent serum specimen.
  3. Patient has malignancy or history of malignancy, with the exception of adequately treated localised squamous cell or basal cell carcinoma, without recurrence.
  4. Patient has been included in another clinical trial protocol for any investigational drug within 4 weeks prior inclusion in UCL-HIA-002.
  5. Patient has any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Inflammatory/immunological reaction and insulin production | 2 years

SECONDARY OUTCOMES:
- Encapsulated human islets function and biocompatibility | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Denis Dufrane, MD, PhD, Principal Investigator — University clinical hospital Saint-Luc
Locations (1):
- University clinical Hospital Saint-Luc, Brussels, Belgium